CLINICAL TRIAL: NCT06115382
Title: Sing for Your Saunter: Using Self-Generated Rhythmic Cues to Enhance Gait in Parkinson's
Brief Title: Sing For Your Saunter Part 2 R33
Acronym: SFYS2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Gammon M Earhart, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202309088
Record Dates: First submitted 2023-09-18; First posted 2023-11-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self cueing (Experimental): Self-cueing training using singing, one hour sessions twice weekly for 12 weeks.
  Interventions: Behavioral: Self Cueing Training
- External cueing (Experimental): External cueing using music, one hour sessions twice weekly for 12 weeks.
  Interventions: Behavioral: External Cueing Training

INTERVENTIONS:
Behavioral: Self Cueing Training — Group classes led by a music therapist and using singing as a self-generated cue, with a focus on rhythm perception, rhythm generation and synchronization of movement to rhythms.
  Arms: Self cueing
Behavioral: External Cueing Training — Group classes led by a music therapist and using music as an external cue, with a focus on rhythm perception, rhythm generation and synchronization of movement to rhythms.
  Arms: External cueing

SUMMARY:
The goal of this clinical trial is to compare to rhythm-based walking interventions to enhance gait in people with Parkinson's disease. The main questions it aims to answer are:

* How does rhythm-based training influence walking performance?
* How does brain activity change following rhythm-based training? Participants will perform walking to music and walking while singing, and will train on the use of these rhythms for 12 weeks. The investigators will compare the effects of training with music to training with singing.

ELIGIBILITY:
Inclusion Criteria:

1. at least 30 years of age
2. diagnosis of idiopathic, typical Parkinson disease according to the UK Brain Bank Criteria
3. Hoehn & Yahr stages 2-3 (mild to moderate disease severity)
4. evidence of walking impairment (score at least 1 on gait item of MDS_UPDRS)

4) stable on all Parkinson disease medications for at least 2 months prior to study entry 5) willing and able to provide informed consent 6) right-handed

Exclusion Criteria:

1. diagnosis of any other neurological condition
2. a score of 2 or greater on item # 3 on the freezing of gait questionnaire
3. significant cognitive impairment
4. unstable medical or concomitant illnesses or psychiatric conditions which, in the opinion of the investigators, would preclude successful participation
5. cardiac problems that interfere with ability to safely participate
6. orthopedic problems in the lower extremities or spine that may limit walking
7. contraindications for magnetic resonance imaging
8. unable to walk for 10 continuous minutes independently
9. left-handed
10. uncontrolled tremor or dyskinesia

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait speed | Baseline and 12 weeks
  How quickly someone walks
MRI Bold Beta Weights | Baseline and 12 weeks
  Measure of blood oxygen levels in different brain regions indicative of level of activity within different brain regions

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Data for individual participants available by request. Only de-identified data will be shared and only for individuals who consent to have their data shared with people who are not part of the original research team.